CLINICAL TRIAL: NCT00384319
Title: Pilot Clinical Study of the LRS ThermoSuit™ System in Post Arrest Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Recovery Systems (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Robert Schock/Vice President Research and Development, Life Recovery Systems
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LRS-01-06-01
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Cardiac Arrest; Comatose
Keywords: resuscitation; hypothermia
MeSH Terms: conditions — Heart Arrest; Coma; Hypothermia | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ThermoSuit(R) System — The ThermoSuit device is used to cool patients using direct contact of the skin with cold water.

SUMMARY:
The purpose of this study is to determine if the Life Recovery Systems Thermosuit(R) System is able to quickly and conveniently cool patients who are comatose after resuscitation from cardiac arrest.

DETAILED DESCRIPTION:
The primary purpose of this study is to clinically evaluate the use of a new cooling device (the LRS ThermoSuit(R) System) to cool patients who are comatose following resuscitation from cardiac arrest. This device cools by circulating cold water directly against the skin of the patient. Cooling to a state of mild hypothermia (32 to 34 degrees C, maintained for 12 to 24 hours) is recognized by the American Heart Association, European Resuscitation Council, and the Canadian Association of Emergency Care Physicians as a promising therapy for such patients, and is likely to be most effective if administered quickly following resuscitation. It is hypothesized that this new device will cool patients much more quickly than by historical means. Patients will be monitored for physiologic parameters such as body temperature during the cooling therapy, and will be tracked for neurological outcomes following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest prior to or during hospital admission, with restoration/return of spontaneous circulation (ROSC).
* Initial (pre-resuscitation) cardiac rhythm of ventricular fibrillation, non-perfusing ventricular tachycardia, pulseless electrical activity, or asystole.
* Estimated or known age > 18 years.
* Intubation, ventilation and placement of esophageal probe.
* Persistent neurologic dysfunction i.e. comatose upon enrollment [GCS ≤ 8].

Exclusion Criteria:

* Height greater than 188 cm.
* Elbow-to-elbow width greater than 60 cm (as measured above the supine patient).
* Core temperature less than 35°C after ROSC (as measured at the tympanic membrane, esophagus, sub-lingual space,nasopharynx, or central blood vessel).
* Comatose state before the cardiac arrest due to the administration of drugs that depress the central nervous system.
* Known pregnancy.
* Response to verbal commands after ROSC (but before enrollment).
* Known terminal illness that preceded the arrest.
* Known enrollment in another study of a device, drug, or biologic.
* Major trauma or other co-morbidity requiring urgent surgery.
* Improving neurologic status.
* > 4 hours since return of spontaneous circulation.
* Unknown time of arrest.
* Severe or known coagulopathy (with active bleeding).
* Hemodynamic instability despite vasopressors (SBP < 90 mmHg or MAP < 60 mmHg for > 30 minutes after ROSC and before enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Primary: Time from collapse to achieving desired range of cooling (32.0 to 34.0°C); | Day of treatment
Time from deployment of the ThermoSuit™ (start of cooled water flow to patient) to core temperature < 34.0°C; | Day of treatment
Total time during the first 24 hours after cooling is initiated that the core temperature is between 32.0 and 34.0°C.; | First day after treatment
Protocol compliance: This is defined as the proportion of patients in whom compliance (i.e. target temperature range) is achieved 85% of the time.; | First day after treatment
Ease of use of the TSS (evaluated by clinical staff using the Product Performance Assessment questionnaire, Appendix 7); | Day of treatment
Duration of maintenance of hypothermia without supplemental cooling; | First day after treatment
Ease of maintenance of hypothermia for 12 hours (whether or not supplemental cooling is needed) | First 12 hours after treatment

SECONDARY OUTCOMES:
Secondary: Total number of days in ICU; | Time while patient is in ICU
Barriers to compliance; | First day after treatment
Neurologic and physical status during in-hospital recovery; | Time while patient is hospitalized
Neurologic and physical status at discharge; | Time at which patient is discharged for hospital
Neurologic and physical status at 30 ± 7 days follow-up for surviving patients; | 30 ± 7 days after hospital discharge
Neurologic and physical status at 6 month ± 15 days follow-up. | 6 months ± 15 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holzer, MD, Principal Investigator — General Hospital, University of Vienna
Locations (1):
- General Hospital, University of Vienna, Vienna, Austria